CLINICAL TRIAL: NCT06285175
Title: REINVENT: A Brain and Muscle Computer Interface for People With Severe Stroke
Brief Title: REINVENT: A Brain and Muscle Computer Interface for Stroke
Acronym: REINVENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Sook-Lei Liew, Associate Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APP-22-04497
Record Dates: First submitted 2022-09-28; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tele-REINVENT (Experimental): All participants in this study are asked to use tele-REINVENT, a 6 week home tele-rehab program with EMG biofeedback.
  Interventions: Other: Tele-REINVENT

INTERVENTIONS:
Other: Tele-REINVENT — Tele-REINVENT consists of EMG-biofeedback of the affected arm to control games on a computer screen.

SUMMARY:
Stroke is a leading cause of adult disability in the United States. High doses of repeated task-specific practice have shown promising results in restoring upper limb function in chronic stroke (>6 months after onset). However, it is currently challenging to provide such doses in standard clinical practice. At-home telerehabilitation services supervised by a clinician are a potential solution to provide higher-dose interventions. However, telerehabilitation systems developed for repeated task-specific practice typically require a minimum level of active movement. Therefore, severely impaired people necessitate alternative therapeutic approaches. Measurement and feedback of electrical muscle activity via electromyography (EMG) have been previously implemented in the presence of minimal or no volitional movement to improve motor performance in people with stroke. Specifically, muscle neurofeedback training to reduce unintended co-contractions of the impaired hand may be a targeted intervention to improve motor control in severely impaired populations. In this study, we examine the effects of a low-cost, portable, and modular EMG biofeedback system (Tele-REINVENT) for supervised and unsupervised upper limb telerehabilitation after stroke during a 6-week home-based training program that reinforces activity of the wrist extensor muscles while avoiding coactivation of flexor muscles via computer games.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe upper extremity hemiparesis and residual hand function (e.g., less than 20 degrees of active wrist or finger extension and enough muscle activity to measure with electromyography).

Exclusion Criteria:

* Taking anti-spasticity medication
* Significant vision loss (corrected vision is acceptable)
* Receptive aphasia
* Hand contractures
* Secondary neurological disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Fugl Meyer Assessment - Upper Extremity | Through study completion, an average of 1 month
  This assessment measures upper limb impairment after stroke
Maximum EMG activity | Through study completion, an average of 1 month
  This assessment measures trace muscle activity in the affected limb during a controlled movement task
Corticomuscular coherence | Through study completion, an average of 1 month
  This assessment measures the connectivity between the brain and muscles of the affected side as a percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No